CLINICAL TRIAL: NCT00003878
Title: The Treatment of One or Two Supratentorial Brain Metastases With Surgical Resection and BCNU-Polymer Wafers
Brief Title: Carmustine Implants in Treating Patients With Brain Metastases
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: New Approaches to Brain Tumor Therapy Consortium (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000067044; NABTT-9802; JHOC-NABTT-9802
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2013-06-21 (Estimated); Status verified 2003-07

CONDITIONS: Metastatic Cancer; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific; tumors metastatic to brain
MeSH Terms: conditions — Neoplasm Metastasis; Brain Neoplasms | interventions — Carmustine

INTERVENTIONS:
Drug: polifeprosan 20 with carmustine implant
Procedure: conventional surgery

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Giving the drugs in different ways may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of implanted carmustine wafers in treating patients who have brain metastases and who are undergoing surgery to remove the tumor.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the local recurrence rate in patients with supratentorial metastatic brain tumors undergoing surgical resection treated with polifeprosan 20 with carmustine implant (Gliadel wafers).
* Determine the incidence and time to recurrence at distant sites within the CNS in these patients after this treatment.
* Determine the median, 6-month, 1-year, and 2-year survival of these patients on this regimen.
* Determine the incidence and severity of cognitive function loss of these patients on this regimen.
* Determine the incidence and severity of CNS and systemic toxic effects of these patients on this regimen.

OUTLINE: Patients receive up to 8 polifeprosan 20 with carmustine implants (Gliadel wafers) implanted in the resected tumor cavity.

Patients are followed on day 7 or day of discharge, at 1 month, 3 months, every 3 months for 21 months, and then for survival.

PROJECTED ACCRUAL: A total of 90 patients will be accrued for this study within 30 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Supratentorial brain metastases for which surgery is recommended

  * Solitary, unilateral, intracranial mass consistent with metastasis on MRI scan OR
  * Two brain lesions consistent with metastases on MRI scan
  * Lesions must be accessible through a single craniotomy
  * Metastatic lesions clearly distinct from tumor bed of any benign lesions
  * Intraoperative frozen section diagnosis of metastatic tumor from CNS lesion
* No prior malignant intracranial neoplasm
* No lesion(s) in the brainstem
* No open communication of the resection cavity with the ventricle following resection

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* Karnofsky 60-100%

Life expectancy

* At least 3 months

Hematopoietic

* No concurrent hematologic disorders

Hepatic

* No concurrent hepatic disease

Renal

* No concurrent renal disease

Cardiovascular

* No concurrent cardiac disease

Pulmonary

* No concurrent pulmonary disorders

Other

* Not pregnant or nursing
* Fertile patients must use effective contraception
* Mini mental score at least 15
* No known hypersensitivity to carmustine or Gliadel wafers
* No other serious concurrent medical illness or infection

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* Not specified

Endocrine therapy

* Not specified

Radiotherapy

* No prior cranial irradiation

Surgery

* See Disease Characteristics
* No prior surgery involving brain metastases or primary brain tumor(s) (except for benign intracranial lesions such as pituitary adenoma, meningioma, or schwannoma)

Other

* Concurrent systemic therapy allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2002-04; Study Completion 2003-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro Olivi, MD, Study Chair — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (11):
- United States (11):
  - University of Alabama at Birmingham Comprehensive Cancer Center, Birmingham, Alabama
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Emory University Hospital - Atlanta, Atlanta, Georgia
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - Lineberger Comprehensive Cancer Center, UNC, Chapel Hill, North Carolina
  - Comprehensive Cancer Center at Wake Forest University, Winston-Salem, North Carolina
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - University of Pennsylvania Cancer Center, Philadelphia, Pennsylvania
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas